CLINICAL TRIAL: NCT06127706
Title: Second Training vs Naive Performer on Second Twin Delivery on Mannequin
Brief Title: Recognition of Second Twin. Second Training vs Naive Performer. PROMPT Mannequin
Acronym: twin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, Director, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ObGynEASC003
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-10

CONDITIONS: Twin Vaginal Delivery Skills

STUDY DESIGN:
Intervention Model Description: two groups randomized One with previous lecture and training, one without
Who Masked: Participant
Masking Description: the two groups are invited for a lecture and are exposed to training skills
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formal lecture and training (Active Comparator): exposure to single test of skills
  Interventions: Device: twin vaginal delivery simulation
- Digital learning only (Active Comparator): exposure to single test of skill
  Interventions: Device: twin vaginal delivery simulation

INTERVENTIONS:
Device: twin vaginal delivery simulation — skill test after formal lecture and simulation in group 1 and after digital learning only
  Other Names: formal lecture; digital learning

SUMMARY:
Anterior foot identification in second twin delivery Two different population of resident in ObGyn Group 1 previous formal lecture on twin vaginal delivery followed by PROMPT mannequin scenario.

Group 2 naive residents

DETAILED DESCRIPTION:
The present study is addressed to evidential skills in residents with and without previous specific didactical approach to twin vaginal delivery in identification of anterior fetal foot.

The two group are randomized by age, sex, seniority. Both the naive and the previous lecture groups are invited to scenario without knowing the intention to test their skills.

The time to reach, the number of attempts are recorded.

ELIGIBILITY:
Inclusion Criteria:

* residents in Ob Gyn

Exclusion Criteria:

* none

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
time to identify foot | 6 weeks after lecture
  time needed to identify foot
number of attempt to identify foot | 6 weeks after lecture
  number of attempt

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Celentano, Pescara, Italia, Italy

IPD SHARING:
Plan to Share IPD: No
All data record are available in Cloud to investigators only due to privacy.

REFERENCES:
- [Background] Gauthier S, Jeanneteau P, Legendre G, Boulvais E, Collin R, Malo L, Rolland D, Courtin O, Thubert T, Winer N, Dochez V. Vaginal delivery of the second twin: A simulation program for residents in obstetrics and gynecology in a type III university maternity hospital. J Gynecol Obstet Hum Reprod. 2022 Oct;51(8):102434. doi: 10.1016/j.jogoh.2022.102434. Epub 2022 Jun 26. PMID 35768063
- [Background] Desseauve D, Daelemans C, Farin A, Jauvion IBM, Ceccaldi PF; Prise en charge des Accouchements a Risque eT des Urgences Maternelles PARTUM teaching program. Internal podalic version of second twin: Improving feet identification using a simulation model. Eur J Obstet Gynecol Reprod Biol. 2022 Aug;275:9-11. doi: 10.1016/j.ejogrb.2022.05.036. Epub 2022 Jun 6. PMID 35691221
- [Background] Celentano C, Prefumo F, Matarrelli B, Mastracchio J, Mauri S, Rosati M. Comparison of practice vs theory model training for vacuum-assisted delivery: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2023 Nov;290:109-114. doi: 10.1016/j.ejogrb.2023.09.024. Epub 2023 Sep 26. PMID 37776704